CLINICAL TRIAL: NCT05188599
Title: Are There Any Relationship Between Isokinetic Parameters and the Amputee Mobility Predictor Scale?
Brief Title: Isokinetic Parameters and the Amputee Mobility Predictor Scale
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associated Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: Gaziler
Record Dates: First submitted 2021-12-10; First posted 2022-01-12 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Amputation, Traumatic
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amputee patients: age between 18-65 years, (b) time after amputation ≥ 6 months, (c) unilateral or bilateral amputation above the ankle level
  Interventions: Diagnostic Test: İsokinetic assessment

INTERVENTIONS:
Diagnostic Test: İsokinetic assessment — Isokinetic assessments of hip flexor and extensor muscle strength and proprioception wiill be performed

SUMMARY:
There is very limited research examining isokinetic parameters and activity level in patients with amputation.. Therefore, the aims of this study were to illustrate isokinetic measurements including strength and proprioception and to analyze the correlation between those isokinetic parameters and activity level and to predict amputee mobility score. It is hypothesized that muscle strength and proprioception were associated with activity level and could be used to estimate amputee mobility scale score in patients with amputation.

DETAILED DESCRIPTION:
Isokinetic measurements are used in the rehabilitation of amputee patients and to evaluate the effectiveness of rehabilitation. The parameters that are frequently looked at in these measurements are isokinetic muscle strength and proprioception. There is very limited research examining isokinetic parameters and activity level in patients with amputation.. Therefore, the aims of this study were to illustrate isokinetic measurements including strength and proprioception and to analyze the correlation between those isokinetic parameters and activity level and to predict amputee mobility score. We hypothesized that muscle strength and proprioception were associated with activity level and could be used to estimate amputee mobility scale score in patients with amputation

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Time after amputation ≥ 6 months
* Unilateral or bilateral amputation above the ankle level

Exclusion Criteria:

* Upper extremity amputation
* The presence of musculoskeletal or neurological disease that could cause functional impairment other than amputation
* The presence of neurological deficit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 43 patients with lower limb amputations
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Isokinetic muscle strength | Through study completion, an average of 1 month
  Muscle strength will be assessed for flexion and extension of the hip using a computer-assisted isokinetic system (CYBEX) in the isokinetic performance laboratory
Isokinetic proprioception | Through study completion, an average of 1 month
  Isokinetic proprioception will be measured with the CYBEX device. The hip joint is chosen because the most proximal level amputation will be the above-knee level
Amputee mobility predictor | Through study completion, an average of 1 month
  Amputee mobility predictor (AMP) is one of the performance-based outcome measures commonly used prior to prosthetic fitting and predict function following prosthetic prescription.The AMP is a 21-item tool for predicting the level of ambulation by assessing static and dynamic balance, transfers, and gait. With this scale, unilateral patients can be evaluated with or without prosthesis. However, activity level of bilateral amputees can only be predicted if they have prostheses. In this study, AMP evaluation of all patients will be performed by a physiotherapist with 10 years of experience in amputee rehabilitation, blinded to other clinical information.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)